CLINICAL TRIAL: NCT02321618
Title: Barber-Pharmacist Coordination to Improve Blood Pressure Management in Black Men
Brief Title: Cut Your Pressure Too: The Los Angeles Barbershop Blood Pressure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); The California Endowment (Other); University of California, Los Angeles (Other); Lincy Foundation (Other)
Responsible Party: Principal Investigator, Ron Victor, DIRECTOR, CEDARS-SINAI HYPERTENSION CENTER DIRECTOR OF CLINICAL RESEARCH & ASSOCIATE DIRECTOR, HEART INSTITUTE BURNS AND ALLEN CHAIR IN CARDIOLOGY RESEARCH, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00035347; 5R01HL117983-02 (NIH)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure; African American men; Black men; barbershop
MeSH Terms: conditions — Hypertension | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BP measurement & pharmacy (Experimental): BP measurements performed by barber, role model poster exposure in barbershop, and BP medication management visits with study pharmacist
  Interventions: Behavioral: BP measurement & pharmacy
- BP educational materials (Other): Exposure to hypertension educational materials in barbershop
  Interventions: Behavioral: BP educational materials

INTERVENTIONS:
Behavioral: BP measurement & pharmacy — Blood pressure monitoring by barber, blood pressure medication management by pharmacist, role model posters encouraging program participation
  Arms: BP measurement & pharmacy
Behavioral: BP educational materials — Exposure to hypertension educational materials
  Arms: BP educational materials

SUMMARY:
African-American men suffer more than most other groups from hypertension (HTN) but often have less access and less contact with doctors. Previous work by the study's Principal Investigator in Dallas, Texas, and Altadena, California, showed that barbershops are an excellent place to identify black men with high blood pressure and to enlist the aid of their barbers as healthcare extenders.

The purpose of this study in Metro Los Angeles (LA) is to compare two types of barber-based patient-centered blood pressure programs to see which type is more effective in improving the customers' high blood pressure. One type emphasizes blood pressure medication and the other type emphasizes lifestyle modification for high blood pressure.

DETAILED DESCRIPTION:
Uncontrolled hypertension (HTN) is one of the most important causes of premature disability and death among non-Hispanic black men. Indeed, black men have the highest HTN death rate of any U.S. race, ethnic, or gender group, contributing to a lower life expectancy. The age-adjusted HTN-related death rate is 3.3-times higher among black men than white men. To address this major health disparity, the investigators designed a novel community-partnered team approach to improve HTN management among black men and prevent needless strokes, heart attacks, kidney failure, and heart failure.

HTN requires physician (or middle-level provider) interaction to optimize blood pressure (BP) medication; black men have less interaction than black women; and thus far lower rates of HTN treatment (73% vs. 86%) and control (36% vs. 50%). Black-owned barbershops are a uniquely personal setting to discuss health with influential male peers. Barbershop health outreach is well-established, but untested as a vehicle for improving HTN control. Scientific evaluation is crucial to best allocate finite healthcare dollars and avoid promoting a "community health industry" that benefits only the promoters.

Under-treatment of HTN is common in primary care due to competing demands on physicians' time. The best way to improve HTN control is with team-based approaches enlisting pharmacists. They are more accessible than physicians, more knowledgeable about medication, and receive training on patient education. The investigators' new conceptual model links the barber-based intervention to team-based care delivery.

The purpose of this research study is to compare this new conceptual model to another barber-based patient-centered blood pressure program to see which is more effective in improving high blood pressure among Black patrons of African American owned barbershops in LA. Patrons randomized to Group 1 (the new conceptual model) will provide blood pressure readings for patrons aged 35 to 79 years of age and refer those with HTN to a Clinical Pharmacist to work with their doctors in optimizing blood pressure medication.

Patrons of Group 1 shops will also be exposed to role model posters are not intended as recruitment materials, but rather are educational tools that intend to highlight positive experiences of participation. The text of the role model stories will in no way provide statements of the effectiveness of the intervention being evaluated by the present research study. Rather, they are the main health messaging tools needed to promote completion of the program in order to achieve the experiences described. Essentially the document will be used as an intervention tool for peer-based health messaging - stories from real customers in the barbershop modeling target behaviors leading that promote continued participation in the protocol by peers with the hopes of achieving to the detection, treatment, and control of high blood pressure. Each role model story will encourage one of two desired health behaviors of potential subjects with elevated BP: 1) ask the barber to check patients' BP with each haircut, 2) schedule a follow-up visit with the study pharmacist to get patient's blood pressure under control. Large posters in the barbershop will show the model customer, his barber, and the study pharmacist who facilitated the desired behavior change. The model's (participants) own words will be used on the poster.

Group 2 barbershop patrons will be exposed to up-to-date information on high blood pressure and on lifestyle topics for blood pressure and heart health including weight management, healthy cooking, cholesterol lowering, and exercise.

A pre-specified cross-sectional sub study utilized the trial's initial screening population to test for an association between self-reported nocturia (>2 nightly/voids) and elevated daytime (in-barbershop) blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 79 years of age
* Non-Hispanic Black men
* Long-term/frequent barbershop patronage (barbershop patrons having at least one haircut every 6 weeks in the same barbershop for the past 6 months).
* Systolic BP >140 at 2 screenings on 2 separate days
* Complete set of Baseline Data

Exclusion Criteria:

* Women
* Children
* <35 years of age
* Non-black
* Hispanic ethnicity
* New/infrequent patronage (<8 haircuts at same barbershop in last 12 months)
* Systolic BP <140 at either screening
* Currently receiving cancer chemotherapy
* On Dialysis
* Incomplete baseline data
* Serious Plan to Move in the next 1.5 years
* Plans to be out of the area for > 1 month in the next 1.5 years

Ages: 35 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Primary Blood Pressure Outcome - change in systolic blood pressure | 6 months
  The pre-specified primary outcome was the change in systolic blood pressure from baseline to 6 months follow-up.

SECONDARY OUTCOMES:
Secondary Blood Pressure Outcome - change in diastolic blood pressure | 6 months
  The change in diastolic blood pressure from baseline to 6 month follow-up
The percentage of participants achieving blood pressure goal | 6 months
  The percentage of participants who achieved blood pressure goal after 6 months follow-up (140/90,135/85, 130/80)
The change in number/type of drug classes prescribed | 6 months
  The change in number/class of prescription drugs prescribed from baseline to 6 month follow-up
Adverse Drug Reactions | 6 months
  The number and type of adverse drug reactions reported from baseline to 6 month follow-up
Self-Rated Health | 6 months
  The change in self-rated health score from baseline to 6 month follow-up
Self-Rated Patient Engagement | 6 months
  The change in PACIC patient engagement score from baseline to 6 month follow-up

OTHER OUTCOMES:
Extension Study Primary Blood Pressure Outcome - change in systolic blood pressure | 12 months
  The primary outcome of the extension study is the change in systolic blood pressure from baseline to 12 months follow-up.
Extension Study Secondary Blood Pressure Outcome - change in diastolic blood pressure | 12 months
  The change in diastolic blood pressure from baseline to 12 month follow-up
Extension Study Secondary Outcome - the percentage of participants achieving blood pressure goal | 12 months
  The percentage of participants who achieved blood pressure goal after 12 months follow-up (140/90,135/85, 130/80)
Extension Study Secondary Outcome - the change in number/type of drug classes prescribed | 12 months
  The change in number/class of prescription drugs prescribed from baseline to 12 month follow-up
Extension Study Secondary Outcome - adverse drug reactions | 12 months
  The number and type of adverse drug reactions reported from baseline to 12 month follow-up
Extension Study Secondary Outcome - self-rated health | 12 months
  The change in self-rated health from baseline to 12 month follow-up
Extension Study Secondary Outcome - self-rated patient engagement | 12 months
  The change in PACIC patient engagement score from baseline to 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Victor RG, Li N, Blyler CA, Mason OR, Chang LC, Moy NPB, Rashid MA, Weiss JP, Handler J, Brettler JW, Sagisi MB, Rader F, Elashoff RM. Nocturia as an Unrecognized Symptom of Uncontrolled Hypertension in Black Men Aged 35 to 49 Years. J Am Heart Assoc. 2019 Mar 5;8(5):e010794. doi: 10.1161/JAHA.118.010794. PMID 30827133
- [Derived] Victor RG, Blyler CA, Li N, Lynch K, Moy NB, Rashid M, Chang LC, Handler J, Brettler J, Rader F, Elashoff RM. Sustainability of Blood Pressure Reduction in Black Barbershops. Circulation. 2019 Jan 2;139(1):10-19. doi: 10.1161/CIRCULATIONAHA.118.038165. PMID 30592662
- [Derived] Victor RG, Lynch K, Li N, Blyler C, Muhammad E, Handler J, Brettler J, Rashid M, Hsu B, Foxx-Drew D, Moy N, Reid AE, Elashoff RM. A Cluster-Randomized Trial of Blood-Pressure Reduction in Black Barbershops. N Engl J Med. 2018 Apr 5;378(14):1291-1301. doi: 10.1056/NEJMoa1717250. Epub 2018 Mar 12. PMID 29527973